CLINICAL TRIAL: NCT03205865
Title: Natural History of Pre-Diabetic Autoimmunity
Brief Title: Diabetes Autoimmunity Study in the Young
Acronym: DAISY
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 92-080
Record Dates: First submitted 2017-06-08; First posted 2017-07-02 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological samples collected at one or more clinic visits include: whole blood, serum, plasma, red blood cells, white blood cells (buffy coat), throat swab, rectal swab, urine, saliva.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Type 1 diabetes (T1D) affects 1.4 million people in the U.S. and its incidence has doubled over the past 20 years. The Diabetes Autoimmunity in the Young Study (DAISY) will estimate overall burden of T1D and other autoimmune diseases in the general population by age 30. The study will evaluate environmental risk factors for development of islet autoimmunity and progression to T1D.

DETAILED DESCRIPTION:
Children determined to be at an increased risk for development of type 1 diabetes, either due to known genetic markers or due to family history of T1D, are followed from birth and monitored for development of T1D-related autoimmunity, on an annual basis. At annual clinic visits, participants are tested for development of these autoantibodies and data is collected related to environmental exposures. In addition to blood collection for determination of autoantibodies, serum and plasma are frozen, and stored for future analyses. Other biological samples collected for further future analysis include: throat swabs, rectal swabs, saliva, and urine. If T1D-related autoantibodies are detected, the participant is asked to increase the frequency of clinic visits to 2-4 visits per year in order to more closely monitor for onset of disease. The endpoint of the study is diagnosis of T1D per the American Diabetes Association (ADA) criteria.

ELIGIBILITY:
Inclusion Criteria:

General Population Genetic Screening to determine Enrollment Eligibility for the Follow-Up Study Criteria

* Child born at St. Joseph Hospital between 1/1/1993 and 6/30/2006
* Informed consent for genetic screening obtained
* Cord blood sample available
* No other severe co-existent condition
* At least one parent/guardian speaks English

General Population Follow Up Study Criteria

* Informed consent for Follow Up obtained
* Initial telephone interview at 3 months of age, initial blood draw at 9 months of age
* High or moderate risk of T1D, as determined from genetic screening (300 low risk children also enrolled as a control group)

Sibling/offspring Follow Up Criteria

* Informed consent for follow up obtained
* Age < 4 yrs (< 7 yrs prior to 1997)
* No other severe co-existent condition
* At least one parent/guardian speaks English

Family Members Follow Up Criteria

* Informed consent obtained
* First degree relative of either a sibling/offspring participant or general population newborn participant
* No other severe co-existent condition
* Ages 12 months to 65 years
* One clinic visit to obtain blood for genetic marker determination and islet autoantibody screening

TEDDY Grad participants

* Completed the TEDDY protocol
* TEDDY home center is Colorado, Washington, Georgia
* Upon completion of the TEDDY protocol, persistently positive for islet autoantibodies at 13.5 yrs of age or older
* Not diagnosed with T1D
* Informed Consent obtained

Exclusion Criteria:

* Cord blood was not available for genetic screening,
* Other severe co-morbidities were indicated,
* Parents refused consent to screening or follow-up,
* At least one parent or legal guardian did not speak English, or
* If T1D had been diagnosed.

Individuals were not eligible to be enrolled into the DAISY study under the Sibling/offspring criteria if:

* They did not have a first degree relative with T1D,
* Other severe co-morbidities were indicated,
* They were older than 4 years of age (older than 7 years of age, before 1997),
* Parents refused consent to follow-up,
* At least one parent or legal guardian did not speak English, or
* T1D had been diagnosed.
* Individuals do not agree to the long-term storage of data and specimen samples.

Ages: 1 Month to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population was selected from among the eligible population in the Denver Metropolitan are as described in the section above. Approximately 50% of the participants are female. The ethnic distribution in the general population newborn cohort is representative of the general Denver Metro area population: 7% African American, 30% Hispanic, 56% non-Hispanic white, and the remaining of biracial or other ethnicity. The ethnic distribution of the sibling/offspring cohort is representative of T1D in the general U.S. population: 5% African American, 10% Hispanic and 85% non-Hispanic white.
Sampling Method: Non-Probability Sample
Enrollment: 2700 (Estimated)
Dates: Start 1993-12-06 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Type 1 Diabetes | From date of birth until the date of first documentation of type 1 diabetes up to 30 years of age.
  Children determined to be at an increased risk for development of type 1 diabetes (T1D), either due to known genetic markers or due to family history of T1D, are followed from birth and monitored for development of T1D-related autoimmunity, on an annual basis. The endpoint of the study is diagnosis of T1D per the American Diabetes Association (ADA) criteria.

SECONDARY OUTCOMES:
Detection of Islet Autoantibodies | From date of birth until the date of first documentation of Islet auto-antibodies up to 20years of age.
  At annual clinic visits, participants are tested for development of these auto-antibodies and data is collected related to environmental exposures. In addition to blood collection for determination of auto-antibodies, serum and plasma are frozen, and stored for future analyses.

OTHER OUTCOMES:
Detection of Transglutaminase Antibodies | From date of birth until the date of first documentation of Transglutaminase auto-antibodies up to 18 years of age.
  At annual clinic visits, using a validated assay, detection of a Celiac Disease related antibody, transglutaminase indicates seroconversion and isolates a period of time in which a change in the immune response, targeting the small intestine.

CONTACTS AND LOCATIONS:
Overall Officials: Marian J Rewers, MD, PhD, MPH, Principal Investigator — Executive Director-Barbara Davis Center for Diabetes, Professor

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available through the National Institute of Diabetes and Digestive and Kidney Disease (NIDDK) repository following manuscript publication which includes such data in the analysis.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available by February 29, 2020. There will not be a limit on the duration of the availability of the data.
Access Criteria: All requests for access of these data sets must be submitted through written request to the PI, Dr. Marian Rewers. Access for the data will be determined by the PI, Dr. Marian Rewers. All investigators who receive DAISY resources must agree to acknowledge the DAISY Study and all co-investigators. This approach is fully compliant with the NIH public data sharing policy.